"Evaluation of the Effect of Life with food allergies education Based on Pender's health Promotion Model Given face to face oath via Social Media to parents of children with food Allergies "

**INFORMED CONSENT FORM** 

Number:.....

04.08.2024

### INFORMED CONSENT FORM

#### PLEASE TAKE THE TIME TO READ THIS DOCUMENT CAREFULLY

Evaluation of the Effect of Life with Food Allergies Education Based on Pender's Health Promotion Model Given Face to Face and via Social Media to Parents of Children with Food Allergies " conducted by Ayşe ÖZEFLANİLİ to the research titled We invite you. Before you decide whether or not to participate in this research, you need to know why and how the research will be conducted. Therefore, it is of great importance to read and understand this form. If there are things you do not understand or are not clear to you, or if you would like more information, ask us.

Participating in this study is entirely <u>voluntary</u>. Not <u>participating</u> in the study or <u>withdrawing</u> from the study at any time after participating You have about. <u>By responding to the study</u>, <u>you are giving your consent to participate in the research</u>. It will be interpreted as . Do not be under anyone's pressure or suggestion when answering the questions <u>on the forms</u> given to you . The information obtained from these forms will be used entirely for research purposes.

### 1. Information about the research:

- a. Purpose of the Research: It will be ensured that the knowledge level, symptom management levels of food allergies, and treatment knowledge levels of parents of children diagnosed with food allergies will be increased.
- b. Content of the Research: Raising awareness of parents by providing Life with Food Allergy Education face to face and via social media, and applying a data collection form.
- c. Reason for Research: Thesis study
- d. Estimated Duration of the Research: 3 weeks
- e. Number of Participants/Volunteers Expected to Participate in the Research: **52**
- f. Place( s ) where the research will be conducted: Kastamonu Training and Research Hospital

## 2. Consent to Participate in the Study:

I have read the above information that must be given to the participant/volunteer before the research, and I fully understand the scope and purpose of the study in which I am asked to participate and my responsibilities as a volunteer. Written and verbal explanations about the study were made by the researcher named below, I had the opportunity to ask questions and discuss and received satisfactory answers. The possible risks and benefits of the study were also explained to me verbally. I understood that I could quit this study whenever I wanted and without having to give any reason, and that I would not face any negative consequences if I quit.

Under these circumstances, I agree to participate in this research voluntarily, without any pressure or coercion.

| Participant (in his/her own handwriting) Name and surname: |
|---|
| Signature: |
| (If any) For Those Under Guardianship or Guardianship; Parent or Guardian (in own handwriting) Name and surname: |

# Signature:

**Note:** This form is issued in two copies. One of these copies is given to the volunteer in return for signature, and the other is kept by the researcher.